CLINICAL TRIAL: NCT04424277
Title: Deformation of the Diaphragm Zone of Apposition During the Loading of the Respiratory System in the Healthy Volunteer. Evaluation of a New Index Measured by Speckle Tracking
Brief Title: Deformation of the Diaphragm Zone of Apposition
Acronym: ZADSPECTRA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: ZADSPECTRA
Record Dates: First submitted 2019-07-22; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2019-10

CONDITIONS: Respiratory Physiology
Keywords: diaphragm; ultrasound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: diaphragm ultrasound — respiratory loading

SUMMARY:
The assessment of the work of the respiratory muscles is a fundamental clinical data in intensive care, especially to guide the management of patients requiring ventilatory support. This data is difficult to access in current practice. The reference technique to estimate the work of breathing (transdiaphragmatic pressure) is not feasible in clinical routine and evaluates only the respiratory work of the diaphragm, not that of the accessory muscles. The ultrasound technique of speckle tracking allows a fine and multidimensional analysis of the deformation of the respiratory muscles during the respiratory cycle.

The investigators hypothesize that the analysis of the multidimensional deformation of the diaphragm at the level of the apposition zone can produce a robust and reproducible index, which is correlated with the work of breathing. The performance of this index will be compared to that of the thickening fraction of the diaphragm. On the other hand, the investigators will evaluate the feasibility of measuring the thickening of the accessory respiratory muscles (scalene and intercostal).

DETAILED DESCRIPTION:
Fifteen healthy subjects will be equipped with a double-balloon esophagogastric tube and subjected to increasing and gradual loading of the respiratory system by a negative-pressure inspiration device. The respiratory work will be recorded continuously by measuring the transdiaphragmatic pressure (reference technique).

The recording of the deformation of the diaphragmatic apposition zone by speckle tracking technique will make it possible to define a multi-dimensional deformation index of this muscular portion.

The reproducibility and the repeatability of this index will be evaluated then this index will be compared to the reference technique, as well as to the fraction of thickening. The deformation of the accessory muscles will also be evaluated in a second step.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer (male or female)
* Free and informed consent

Exclusion Criteria:

* known pregnancy, parturient or nursing mother
* Under 18 years old
* Age> 45 years
* Incapable major
* Non-affiliation to the social security system
* Any history of respiratory pathology
* Any history of coagulation disorder or platelet function

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The subjects and participants will be contacted individually by the investigators. The principles of the study will be explained and explained to the volunteer.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Coefficient of reproducibility | 1 hour
  reproducibility and repetability measurments of strain (ε) and strain rate (ε') .

SECONDARY OUTCOMES:
agreement between the strain and pressure time product of diaphragm (PTPdi) | 1 hour
  Correlation between the strain and pressure time product of diaphragm (PTPdi)
agreement between the strain rate of the PTPdi | 1 hour
  Correlation between the strain rate of the PTPdi
comparison of repeatability and reproducibility of the various ultrasound indices (TEE, TFdi, ε and ε '). | 1 hour
  Comparison of repeatability and reproducibility of the various ultrasound indices (TEE, TFdi, ε and ε ').
Repeatability and reproducibility of the measurement of the deformation (ε) and the rate of deformation (ε ') of the accessory muscles (scalene then intercostal) subjected to variable inspiratory loads. | 1 hour
  Repeatability and reproducibility of the measurement of the deformation (ε) and the rate of deformation (ε ') of the accessory muscles (scalene then intercostal) subjected to variable inspiratory loads.
Exploration of the link between the deformation of the accessory respiratory muscles by speckle tracking and the PTPdi | 1 hour
  Coorelatin between strain of the accessory respiratory muscles and the PTPdi

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe CARMAS, Créteil, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No